CLINICAL TRIAL: NCT05854407
Title: MRI Exploration of Protein Digestion - a Feasibility Study
Brief Title: MRI Exploration of Protein Digestion
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Paul Smeets, Principle Investigator, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL83133.091.23
Record Dates: First submitted 2023-04-19; First posted 2023-05-11 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Gastric Digestion

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pasteurized skim milk (Other): 300 mL of commercial pasteurized skim milk (heated for 15s at ~72 °C)
  Interventions: Other: skim milk
- High-pasteurized skim milk (Other): 300 mL of High-pasteurized skim milk prepared by heating commercial pasteurized skim milk for 30 min at 80 °C
  Interventions: Other: skim milk

INTERVENTIONS:
Other: skim milk — pasteurized or high-pasteurized skim milk

SUMMARY:
The goal of this study is to assess the feasibility of using MRI for in vivo monitoring of gastric milk digestion (protein coagulation and breakdown). The study will be in healthy normal-weight individuals aged between 18 and 45 years.

The main questions it aims to answer are:

1. Is there a significant effect of time on the postprandial magnetization transfer ratio (MTR) of the stomach contents?
2. Can a difference in postprandial MTR of the stomach contents between the test products be detected?

Participants will visit after an overnight fast two times and then have MRI scans of the stomach before and after the consumption of 500 mL of pasteurized or high-pasteurized skim milk.

DETAILED DESCRIPTION:
Rationale: Gastric digestion is the first step in the breakdown of dietary proteins, and is therefore essential for the further breakdown in the intestines and subsequent absorption of amino acids. Food processing, such as heating can modify the structure and digestibility of proteins. Digestion of dietary protein, and how this is affected by heating is often studied using in vitro digestion models that mimic the digestive tract. However, outcomes from these models need to be verified using in vivo digestion data from humans. Such data can in turn be used to improve digestion models. Magnetic resonance imaging (MRI) may be used to non-invasively monitor both in vitro and in vivo protein digestion, and hence, may bridge the gap between in vitro digestion models and real-life digestion physiology. The investigators have recently established candidate MRI markers for gastric protein digestion using in vitro models (MT and CEST MRI). As a next step, their potential for in vivo application needs to be established. Therefore, the aim of this research is to do a feasibility study in humans.

Objective: Assess the feasibility of using MT MRI for in vivo monitoring of gastric milk digestion (protein coagulation and breakdown).

Study design: Randomized cross-over study with two treatments.

Study population: 12 healthy volunteers, 18-45 years old.

Intervention: Participants will ingest 300 mL of commercial pasteurized skim milk (SM, heated for 20 s at 72 °C) and of high pasteurized skim milk (heated for 30 min at 80 °C). MRI scans of the stomach will be made at baseline, at t = 5 min and at 15-minute intervals up until t = 95 minutes after the start of ingestion. In addition, verbal ratings of hunger, fullness and nausea will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45y
* Apparently healthy
* Normal weight (BMI 18.5-25)

Exclusion Criteria:

* Milk protein allergy or intolerance (self-reported)
* Lactose intolerance (self-reported)
* Gastric disorders or regular (>once a week) gastric complaints such as heartburn
* Use of medication which alters the normal functioning of the stomach, such as:

  * medical drug use that influences the GI tract's normal function, e.g. motility, and pH. For example, proton pump inhibitors, antacids, anti-depressants etc. (judged by our study doctor)
* Use of recreational drugs within one week before the test day (marihuana, XTC, GHB, helium)
* Being pregnant, lactating or planning on becoming pregnant during the study
* Alcohol consumption of more than 7 glasses per week
* Smoking (>2 cigarettes a week)
* Having gained or lost more than 5 kg of weight in the last month.
* Participating in other biomedical research during the study period
* Having a contra-indication to MRI scanning:

  * Intraorbital or intraocular metallic fragments
  * Ferromagnetic implants
  * Claustrophobia (self-reported)
* Unwillingness to be referred to their general practitioner in case of chance findings of pathology
* Being an employee or student of the Division of Human Nutrition and Health or the Laboratory of Biophysics at Wageningen University.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
MT MRI scans of the stomach | Baseline, T = 5, 20, 35, 50, 65, 80, 95 minutes after start of consumption
  average MTR of the stomach content over time

SECONDARY OUTCOMES:
CEST MRI of the stomach | Baseline, T = 5, 20, 35, 50, 65, 80, 95 minutes after start of consumption
  Average CESTR of the stomach content over time (measure of soluble proteins and peptides)

OTHER OUTCOMES:
Verbal subjective ratings of appetite, thirst and wellbeing provided on a scale of 0 - 100 units | Baseline, T = 5, 20, 35, 50, 65, 80, 95 minutes after start of consumption
Gastric content volume | Baseline, T = 5, 20, 35, 50, 65, 80, 95 minutes after start of consumption
  Change from baseline gastric content volume over time in milliliter as determined from an abdominal MRI scan

CONTACTS AND LOCATIONS:
Locations (1):
- Human Research Unit - Division of Human Nutrition and Health, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No